CLINICAL TRIAL: NCT03147924
Title: Examining the Effects of an Improvisation Group on Social Anxiety Among Help-seeking Youth
Brief Title: Examining the Effects of an Improvisation Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Juliana Tobon, Psychologist, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2927
Record Dates: First submitted 2017-05-03; First posted 2017-05-10 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Anxiety; Depression; Self Concept Alteration; Social Support
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attending Improvisation Group (Experimental): Attended 3 or more Improvisation Group sessions
  Interventions: Other: Improvisation Group

INTERVENTIONS:
Other: Improvisation Group — The aim of this pilot study is to investigate the effects of improvisational comedy in a group of help-seeking youth at risk of developing a range of mental health disorders, including social anxiety.

SUMMARY:
This study is taking place to examine the preliminary effects of improvisational therapy (improv group) on social anxiety for youth at the Youth Wellness Centre (YWC). The improv group will run for 12-weeks as a drop-in group. A typical session will begin with stretching, simple breathing and an activity to promote group cohesion. Following this, improvisation games and activities will be introduced with the goal of promoting the following skills: assertiveness, acceptance, problem solving, co-operate skills, non-verbal communication, mindfulness, and memory. Youth who consent to the study will be asked to complete a set of brief questionnaires the first time they attend one of the sessions. Youth who have attended at least 3 sessions will be asked again to complete questionnaires following the completion of week 12 session. Youth will also rate their anxiety and distress on a simple rating scale at the beginning and end of each session. Additionally, all participants (who have attended three or more sessions) will be invited to complete a 30 to 45 minute qualitative interview following the 12 week session. Participants are predicted to show a decrease in social anxiety, generalized anxiety and depression symptoms, and an increase in self-esteem, and perceived social support.

ELIGIBILITY:
Inclusion Criteria:

* help-seeking youth
* ages 17-25

Exclusion Criteria:

* will NOT be excluded on the basis of mental health or addiction concerns

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder 7 (GAD-7) | Pre-group and 12-weeks later (post group)
  A seven-item self-report anxiety questionnaire designed to monitor and assess the severity of generalized anxiety disorder (GAD) symptoms.
Change in Social Phobia Inventory (SPIN) | Pre-group and 12-weeks later (post group)
  A seventeen-item questionnaire used to measure the severity of social anxiety.
Change in Subjective Units of Distress Scale (SUDS) | Pre and post every improv session for a duration of 12-weeks
  A thermometer scale used to track anxiety before and after each session

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) | Pre-group and 12-weeks later (post group)
  A nine-item questionnaire used to measure depression
Change in Kessler Psychological Distress Scale (K-10) | Pre-group and 12-weeks later (post group)
  A 10-item questionnaire intended to measure distress based on questions about anxiety and depressive symptoms.
Change in Rosenberg Self-Esteem Scale (RSES) | Pre-group and 12-weeks later (post group)
  A 10-item questionnaire used to measure self-esteem.
Change in Multidimensional Scale of Perceived Social Support (MSPSS) | Pre-group and 12-weeks later (post group)
  A 12-item questionnaire designed to measure perception of support from 3 sources: family, friends and significant other

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Tobon, PhD.,C.Psych, Principal Investigator — St. Joseph's Research Institute
Locations (1):
- Youth Wellness Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinsola, E.F., & Udoka, P.A.. Parental Influence on Social Anxiety in Children and Adolescents: Its Assessment and Management Using Psychodrama. Psychology. 4(3A), 246-253, 2013.
- [Background] Albano, A. M. & Kendall, P.C. (2002). Cognitive Behavioural Therapy for Children and Adolescents with Anxiety Disorders: Clinical Research Advances. International Review of Psychiatry, 14, 129-134.
- [Background] Bagley C, Bolitho F, Bertrand L. Norms and Construct Validity of the Rosenberg Self-Esteem Scale in Canadian High School Populations: Implications for counselling. Canadian Journal of Counselling. 1997;31(1):82.
- [Background] Benjamin CL, O'Neil KA, Crawley SA, Beidas RS, Coles M, Kendall PC. Patterns and predictors of subjective units of distress in anxious youth. Behav Cogn Psychother. 2010 Jul;38(4):497-504. doi: 10.1017/S1352465810000287. Epub 2010 May 28. PMID 20509987
- [Background] Bermant G. Working with(out) a net: improvisational theater and enhanced well-being. Front Psychol. 2013 Dec 10;4:929. doi: 10.3389/fpsyg.2013.00929. eCollection 2013. No abstract available. PMID 24339820
- [Background] Besser A, Weinberg M, Zeigler-Hill V, Ataria Y, Neria Y. Humor and Trauma-Related Psychopathology Among Survivors of Terror Attacks and Their Spouses. Psychiatry. 2015;78(4):341-53. doi: 10.1080/00332747.2015.1061312. PMID 26745687
- [Background] Butler, M. & Pang, M. (2014). Current Issues in Mental Health in Canada: Child and Youth Mental Health. Parliamentary Information and Research Service, Library of Parliament, Publication no. 2014-13.
- [Background] Connor KM, Davidson JR, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). New self-rating scale. Br J Psychiatry. 2000 Apr;176:379-86. doi: 10.1192/bjp.176.4.379. PMID 10827888
- [Background] Ferner RE, Aronson JK. Laughter and MIRTH (Methodical Investigation of Risibility, Therapeutic and Harmful): narrative synthesis. BMJ. 2013 Dec 12;347:f7274. doi: 10.1136/bmj.f7274. PMID 24336308
- [Background] Hayes SA, Miller NA, Hope DA, Heimberg RG, Juster HR. Assessing Client Progress Session by Session in the Treatment of Social Anxiety Disorder: The Social Anxiety Session Change Index. Cogn Behav Pract. 2008 May 1;15(2):203-2011. doi: 10.1016/j.cbpra.2007.02.010. PMID 25075171
- [Background] Kendall, P.C., Robin, J.A., Hedtke, K.A., Suveg, C., Flannery-Schroeder, E. & Gosch, E. (2005). Considering CBT with Anxious Youth? Think Exposures. Cognitive and Behavioural Practice, 12, 136-150.
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Kim SH, Kook JR, Kwon M, Son MH, Ahn SD, Kim YH. The effects of laughter therapy on mood state and self-esteem in cancer patients undergoing radiation therapy: a randomized controlled trial. J Altern Complement Med. 2015 Apr;21(4):217-22. doi: 10.1089/acm.2014.0152. PMID 25875938
- [Background] Kindler, R.C. & Gray, A.A. (2010). Theater and Therapy: How Improvisation Informs the Analytic Hour. Psychoanalytic Inquiry, 30, 254-266. doi: 10.1080/07351690903206223
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Mesa F, Beidel DC, Bunnell BE. An examination of psychopathology and daily impairment in adolescents with social anxiety disorder. PLoS One. 2014 Apr 1;9(4):e93668. doi: 10.1371/journal.pone.0093668. eCollection 2014. PMID 24691406
- [Background] Misch DA. A PIECE OF MY MIND. I Feel Witty, Oh So Witty. JAMA. 2016 Jan 26;315(4):345-6. doi: 10.1001/jama.2015.16758. No abstract available. PMID 26813204
- [Background] Palinkas LA. Qualitative and mixed methods in mental health services and implementation research. J Clin Child Adolesc Psychol. 2014;43(6):851-61. doi: 10.1080/15374416.2014.910791. PMID 25350675
- [Background] Rudnick A, Kohn PM, Edwards KR, Podnar D, Caird S, Martin R. Humour-related interventions for people with mental illness: a randomized controlled pilot study. Community Ment Health J. 2014 Aug;50(6):737-42. doi: 10.1007/s10597-013-9685-4. Epub 2013 Dec 12. PMID 24337476
- [Background] Sheesley, A.P., Pfeffer, M. & Barish, B. (2016). Comedic Improv Therapy for the Treatment of Social Anxiety Disorder. Journal of Creativity in Mental Health. 11(2), 157-169. doi: 10.1080/15401383.2016
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Steitzer, C. (2011). The Brilliant Genius: Using Improv Comedy in Social Work Groups. Social Worker with Groups, 34, 270-282. doi: 10.1080/01609513.2011.558830
- [Background] Yorton, T. (2005). Using Improv Methods to Overcome the Fear Factor. Wiley Periodicals. doi: 10.1002/ert.20036